CLINICAL TRIAL: NCT07136363
Title: RESTORE Study R61 Pilot Phase: Recovery and Engagement for Stimulant Users on Re-entry
Brief Title: RESTORE Study R61 Phase: Recovery and Engagement for Stimulant Users on Re-entry
Acronym: RESTORE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Ank Nijhawan, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU20251062
Record Dates: First submitted 2025-07-09; First posted 2025-08-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: HIV; Stimulant Use Disorder; Justice Involved Populations; HIV Prevention
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Arm 1: DynamiCare-plus (Experimental): Patient Navigation (PN) with a smartphone with the DynamiCare mobile contingency management app
  Interventions: Device: DynamiCare; Behavioral: Patient Navigation (PN)
- Arm 2: Enhanced Treatment as Usual (ETAU) (Active Comparator): Patient Navigation (PN) with a smartphone without the DynamiCare app
  Interventions: Behavioral: Patient Navigation (PN)

INTERVENTIONS:
Device: DynamiCare — DynamiCare is a mobile contingency management (CM) platform. Participants randomized to this intervention receive access to the DynamiCare app, an FDA-approved mobile application that delivers CM through features such as at-home saliva drug testing, appointment check-ins, and incentives for healthy behaviors. The app is designed to promote substance use reduction and engagement in care by providing financial rewards for meeting health-related goals. The intervention aims to improve initiation and retention in HIV prevention or treatment (PrEP or ART), reduce stimulant use, and enhance overall health outcomes among justice-involved individuals.
  Arms: Arm 1: DynamiCare-plus
Behavioral: Patient Navigation (PN) — Participants work with a trained patient navigator (PN) who provides individualized support, assists with linkage to medical and social services, and helps address barriers to care. The PN meets with participants weekly during the first month and biweekly thereafter to conduct a comprehensive needs assessment and provide tailored support. This includes assistance with obtaining housing, identification, insurance, transportation, and linkage to health and social services such as HIV prevention or treatment (PrEP/ART), substance use disorder treatment, and other community-based care. The navigation protocol follows established procedures from prior studies (e.g., ACTION). All participants receive a smartphone to support communication and appointment coordination.

SUMMARY:
Justice-involved individuals face disproportionately high rates of stimulant use disorder and HIV, along with disrupted access to HIV treatment and prevention services like ART and PrEP. Contingency management (CM) is the most effective intervention for stimulant use, but its use in justice-involved populations has been limited by logistical and structural barriers. DynamiCare is an FDA-approved mobile app that delivers behavioral CM and has shown promise in reducing stimulant use, but its impact on HIV-related outcomes remains unknown. The RESTORE study (Recovery and Engagement for Stimulant Users on Re-entry) will evaluate whether combining DynamiCare with patient navigation (DynamiCare-plus) improves PrEP/ART initiation and reduces stimulant use among individuals recently released from justice settings. The R61 phase will assess feasibility, acceptability, and preliminary effectiveness among 40 participants. If milestones are met, the R33 phase will scale to a randomized controlled trial with 252 participants to assess effectiveness, implementation, and cost. This scalable, mobile approach has the potential to address a critical gap in care for a highly vulnerable population.

DETAILED DESCRIPTION:
Stimulant use (cocaine/ methamphetamine) has a major impact on HIV transmission and acquisition. Justice-involved individuals are more likely to have stimulant use disorders and be at risk or living with HIV than the general population, face interruptions in HIV treatment (antiretroviral therapy (ART)) and have limited access to HIV pre-exposure prophylaxis (PrEP). There is thus a critical need for effective interventions that reduce stimulant use and potentially improve HIV viral suppression (VS) and PrEP initiation and retention, particularly among justice-involved groups. The most successful treatment for stimulant use disorder to date is contingency management (CM), shown to reduce stimulant use and HIV risk behaviors, though implementation has been limited for justice-involved people due to competing priorities (transportation, housing, probation) and practical challenges of providing CM (frequent drug testing, trained staff, incentive management). DynamiCare is an FDA-approved mobile app that delivers patient-centered behavioral CM and has been shown to reduce biological and self-reported assessments of stimulant and other substance use, however it is unknown if it could improve PrEP/ART initiation for persons with stimulant use disorder at risk or living with HIV. Thus, in response to NIDA RFA-DA-23-008 [Request for Applications (RFA) from the National Institute on Drug Abuse (NIDA)]: Stimulants and HIV, we propose the RESTORE study: Recovery and Engagement for Stimulant Users on Re-entry. Guided by the Exploration Preparation Implementation Sustainment (EPIS) framework, we will assess if the addition of personalized CM via the DynamiCare app to a previously protocolized patient navigator (PN) ("DynamiCare-plus") intervention improves initiation of PrEP/ART and reduces stimulant use. The Specific Aims are: Aim 1 (R61): To conduct a pilot assessment of DynamiCare-plus for persons at risk or living with HIV with DSM-5 (Diagnostic and Statistical Manual of Mental Disorders-5) stimulant use disorders (methamphetamine/cocaine) being released to the community from a closed justice setting (jail/ prison/ justice-mandated substance use program). N=40 adults in Dallas, TX (Texas) and CT (Connecticut) will be randomized 1:1 to DynamiCare-plus compared to enhanced treatment as usual (ETAU) (PN + smartphone) for 6 months to assess acceptability, feasibility and preliminary effectiveness: proportion who (1) initiate PrEP/ART; and (2) achieve/maintain VS (VL < 200 copies/mL) for those with HIV; Aim 2 (R33): The R61 pilot will inform a type 1 hybrid implementation effectiveness randomized controlled trial of DynamiCare-plus v. ETAU among 252 participants with the same eligibility as the R61 to assess the primary outcome of initiation/reinitiation of PrEP/ART followed for 15 months, with a 12 month intervention period. Secondary outcomes include stimulant and other substance use, overdose, PrEP/ART/SUD (Substance Use Disorder) retention, HIV risk behaviors, VS, Quality of life, and recidivism; Aim 2.1: Examine implementation of the intervention. Aim 2.2: Conduct cost analyses of the intervention compared to control. The Dynamicare app is mobile, adaptable and scalable, and combined with PN (DynamiCare-plus) has the potential to have a major impact on HIV treatment and prevention for justice-involved people with stimulant use disorder.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older
* Have a DSM-5 diagnosis of stimulant use disorder (methamphetamine and/or cocaine)
* Be at risk for or living with HIV
* Be transitioning to the community from a closed justice setting, such as:

Jail Prison Justice-mandated residential substance use program

* Be able to provide informed consent
* Be willing and able to use a smartphone app (DynamiCare)

Exclusion Criteria:

* Severe medical or psychiatric disability making participation unsafe
* Unable to provide consent or engage with the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04-06 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants without HIV taking HIV pre-exposure prophylaxis (PrEP) by validated self-report within 6-month intervention period | 6 months
  Number of participants without HIV who report taking PrEP (initiating or re-initiating PrEP) within the 6-month intervention period, as measured by self-report and validated by medical record and pharmacy fill data, divided by all participants without HIV.
Proportion of participants with HIV taking Antiretroviral therapy (ART) by validated self-report within 6-month intervention period | 6 months
  Number of participants with HIV taking ART (initiating or re-initiating ART) within the 6-month intervention period, as measured by self-report and validated by medical record and pharmacy fill data, divided by all participants with HIV.
Proportion of participants with HIV who achieve HIV viral suppression (VS) by blood assay at month 6 of the intervention. | 6 months
  Number of participants with HIV who achieve (at month 6) an HIV viral load of < 200 copies/mL as measured by real-time PCR (Polymerase Chain Reaction) blood test, divided by all participants with HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Ank Nijhawan, MD, Principal Investigator — University of Texas Southwestern Medical Center; Sandra Springer, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - Parkland County Hospital, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
MPIs (Multiple Principle Investigators) will consider de-identified data sharing upon reasonable request from other researchers.